CLINICAL TRIAL: NCT04686877
Title: Safety and Efficacy of Stereotactic Aspiration Plus Urokinase in Deep Intracerebral Hemorrhage Evacuation: a Multicentral Randomized, Controlled, Open-label, Trial
Brief Title: Safety and Efficacy of Stereotactic Aspiration Plus Urokinase in Deep Intracerebral Hemorrhage Evacuation
Acronym: STAPLE-dICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Collaborators: Department of Science and Technology of Fujian province (Unknown); Longyan City First Hospital (Other); Fifth Affiliated Hospital of Zhengzhou University (Unknown); Shanxi Provincial People's Hospital (Other Government); Tangshan Gongren Hospital (Other); Lanzhou University Second Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other); The Second Hospital of Shandong University (Other); Shishi General Hospital (Unknown); Wuping County Hospital (Unknown); Fuqing Municipal Hospital (Unknown); Qingyuan People's Hospital (Other); Jinjiang Municipal Hospital (Unknown); Anxi County Hospital (Unknown); Nanan Hospital (Unknown); MinDong Hospital of Ningde City (Unknown); Affiliated Hospital of Putian University (Unknown); Lianjiang County Hospital (Unknown); Shunchang County Hospital (Unknown); Yulin No.2 Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); The Second Affiliated Hospital of Xiamen Medical College (Unknown); Zhangzhou Municipal Hospital of Fujian Province (Other); Longyan People's Hospital of Fujian Province (Unknown)
Responsible Party: Principal Investigator, De-zhi Kang, Doctor, First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019Y9118
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Treatment of Spontaneous Intracerebral Hemorrhage
Keywords: Deep-Seated Spontaneous Intracerebral Hemorrhage; Stereotactic Aspiration; Urokinase Irrigation; Randomized Controlled Trial; Long-term outcome
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Intervention Model Description: A surgical intervention model of stereotactic hematoma punctural catheter placement, drainage and urokinase irrigation in spontaneous intracerebral hemorrhage.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors assessed the outcome of patients on the basis of follow-up visits by telephone or in the clinic, with no knowledge of group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STAPLE group (Experimental): In patients enrolled in the STAPLE group to receive the stereotactic CTA-guided aspiration and drainage, the surgery is performed within 36 h of symptoms onset. Urokinase injection is determined according to the CT scan 6 h after the surgery. Then the optimal dose of urokinase determined in Step A will be given. On the 1st, 3rd, 5th, and 7th day of post-operation, patients will be re-examined using CT. Conventional craniotomy and hematoma evacuation can be performed when cerebral hernia or rebleeding happened.
  Interventions: Procedure: STAPLE
- Conservative treatment group (No Intervention): Patients in the conservative treatment group are treated routinely in accordance with Guidelines for the Management of Spontaneous Intracerebral Hemorrhage (AHA/ASA, 2015) 9. Hematoma evacuation by craniotomy or decompressive hemicraniectomy is considered in deteriorating patients as a life-saving measure.

INTERVENTIONS:
Procedure: STAPLE — Stereotactic aspiration plus urokinase clot irrigation
  Arms: STAPLE group

SUMMARY:
This is a nationwide, multicenter, open-label, randomized controlled trial of early minimally invasive treatment for deep-seated spontaneous cerebral hemorrhage (dICH). The study consists of 2 steps: the first step is to conduct a dose climbing test to determine the safety and optimal dose of urokinase intra-hematoma irrigation after stereotactic aspiration; the second step is to validate whether stereotactic aspiration plus urokinase irrigation (the optimal dose determined in step one) is superior to conservative treatment in improving long-term outcomes (1 year) in early (within 24h) dICH patients.

DETAILED DESCRIPTION:
Surgical options have been repeatedly evaluated in large multicenter randomized controlled trials that unfortunately have not demonstrated improved outcomes. Recently, MISTIE III study concluded that minimally invasive surgery with thrombolysis was safely adopted by doctors, but did not improve the proportion of patients who achieved a good long-term outcome. However, subgroup analyses of MISTIE cohorts showed that patients with GCS≥9, time from stroke to treatment initiation <36 h, and reduction of ICH to ≤15 mL had a higher likelihood of achieving mRS of 0 to 3. Thus, we designed this study, considering the reality of clinical practice in China and the limitations of previous studies, to determine the optimal dose and safety of urokinase intra-hematoma irrigation, and to validate whether stereotactic aspiration plus urokinase irrigation (STAPLE) is superior to conservative treatment in improving long-term outcomes (1 year) in early (within 24h) dICH patients.

The Part A study aimed to find the safe optimal dose of urokinase by a Utility-based Bayesian optimal interval (U-BOIN) phase I/II design. In this design, the dose-limiting toxicity (DLT) is defined as rebleeding that occurred from the first urokinase injection to 72 h after the last injection. And the effective performance is defined as a hematoma volume <10 ml on CT scan after the last injection as well as the total number of injections not exceeding four. he demographic data, medical history, examination results, complications, treatment, and survival information of the participants are recorded during hospitalization. The participants should go to the outpatient clinic on the 30th day after entering the study, and their CT scan and neurological examination results will be recorded. If the participants died, the time and cause of death will be collected. In the Part B study, eligible patients will be randomized in equal proportions between STAPLE group and conservative treatment group immediately after the pre-surgical CTA. The method of block randomization and stratification control is used. Patients in the STAPLE group receive the stereotactic CTA-guided aspiration and drainage within 36h after symptoms onset, and the injection volume of urokinase was determined according to the results of CT examination at 6 hours after operation. Patients in the conservative treatment group are treated routinely according to the Guidelines for the Management of Spontaneous Intracerebral Hemorrhage (AHA/ASA, 2015). Hematoma evacuation by craniotomy or decompressive hemicraniectomy is considered in deteriorating patients as a life-saving measure. Subjects will be followed up by phone at days 90, 180, and 270. And the survivors should go to the outpatient clinic of the participating centers at day 30 and day 365 after randomization. Their CT results and neurological physical examination (including but not limited to mRS, Glasgow Outcome Score (GOS), and Barthel Index (BI)) will be recorded.

ELIGIBILITY:
Inclusion criteria:

1. aged 40 years or older;
2. the duration from onset to the baseline computed tomography angiography (CTA) scan was between 6 to 24 hours;
3. patients with a spontaneous ICH in the deep brain parenchyma (≥1 cm from the cortical surface); with hematoma volume more than 25 ml (measured with the ABC/2 method); without hydrocephalus caused by intraventricular hemorrhage; without cerebral herniation and the benefit of surgical treatment was unknown;
4. The Glasgow Coma Scale (GCS) ranged from 9 to 15;
5. patients with motor deficits;
6. The modified Rankin Score (mRS) ranged from 0 to1 before onset.

Exclusion Criteria:

1. ICH was caused by aneurysms, arteriovenous malformations, tumors, or trauma;
2. patients had a history of intracerebral hemorrhage or ischemic cerebral infarction;
3. patients had severe coagulation disorders with INR ≥ 1.5;
4. patients had severe underlying diseases, which may affect the outcomes;
5. pregnant and lactating patients;
6. patients refused to sign the informed consent and receive follow-up.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Good functional outcome, measured by the modified Rankin Scale (mRS) | At day 365 after randomization
  Good functional outcome is defined as a mRS of ≤3 points and will be assessed as binary outcome (yes/no, final value). In this context, a mRS score of 3 points reflects the ability to walk unassisted and care for one's own bodily needs despite being moderately dependent on assistance, while a mRS score of 4 points describes a patient who is not able to walk anymore and needs assistance with all daily activities and thus marks a severe loss of patient autonomy.

SECONDARY OUTCOMES:
Proportion of hematoma evacuation by craniotomy or decompressive hemicraniectomy | at 1 year after randomization
  Number of participants who were converted to hematoma evacuation by craniotomy or decompressive hemicraniectomy for reasons such as hematoma enlargement after conservative treatment or urokinase treatment.
Residual hematoma volume | At day 7 after randomization in the Conservative Treatment group; At 72 hours after the last urokinase infusion in the STAPLE group
  Proportion of patients with hematoma volume reduced to less than 10mL [binary outcome (yes/no)]. The hematoma volume will be measured on cranial computer tomography (cCT) at day 7 after randomization in the Conservative Treatment group and 72 hours after the last urokinase infusion in the STAPLE group.
All-cause mortality | At 365 days after randomization
  Mortality rate as measured by death of a participant [binary outcome (yes/no)]. Death induced by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Kang Dezhi, MD., Study Chair — The first affilicated hospital of Fujian Medical univercity
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
We will share individual participant data after the primary results have been published.

REFERENCES:
- [Derived] Yan Z, Jiang L, Li G, Xia K, Peng L, Hu J, Chen S, Zhang J, Huang X. Efficacy study of neuronavigation-assisted stereotactic drilling of urokinase drainage versus craniotomy in the treatment of massive intracerebral haemorrhage in elderly patientsa. Sci Rep. 2024 Sep 3;14(1):20439. doi: 10.1038/s41598-024-71130-x. PMID 39227662